CLINICAL TRIAL: NCT04679792
Title: Postural Control Quality in Chiari I Malformation: Evaluation in a Pediatric Population
Brief Title: Postual Control in Pediatric Chiari I Malformation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other)
Responsible Party: Principal Investigator, Philippe PERRIN, Professor, Central Hospital, Nancy, France
Other Study IDs: EquiChiari
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Chiari I Malformation; Pediatric
MeSH Terms: conditions — Arnold-Chiari Malformation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- operated: Patients Under 18 years of age who are operated for Chiari Malformation on the basis of routine neurosurgical assessment.
  Interventions: Diagnostic Test: Dynamic posturography
- non operated: Patients Under 18 years of age who are not operated for Chiari Malformation on the basis of routine neurosurgical assessment.
  Interventions: Diagnostic Test: Dynamic posturography

INTERVENTIONS:
Diagnostic Test: Dynamic posturography — Balance evaluation

SUMMARY:
BACKGROUND: Chiari I malformation is a rare disease characterized by cerebellar amygdalae descent under the level of the foramen magnum. It causes troubles in cerebrospinal fluid circulation and direct compression on brainstem, producing characteristic headaches, neurological impairment and syringomyelia. Surgery is the only treatment, indicated when symptomatology exists. However, sometimes patients complaint about atypical symptoms that are difficult to interpret.

We would like to study one of these atypical symptoms, gait imbalance, in a pediatric population thanks to a computerized dynamic posturography (Equitest®).

METHOD: infants from 6 to 18 years of age presenting a radiologically confirmed Chiari I malformation will be included in the study. We will compare posturographic results of patients which will be operated on with the results of the patients which will not; furthermore, we will compare preoperative and postoperative results in operated patients.

RESULTS: 19 patients have been enrolled in the study, and data have been collected for 12 of them. Seven patients belong to operated population.

CONCLUSIONS: even if enrolment of the patients is satisfactory, disposable data are not enough to perform statistical analysis and to put forward any conclusion.

DETAILED DESCRIPTION:
Chiari malformation is characterized by at least 5 mm descent of cerebellar tonsils below the foramen magnum, into the vertebral canal. Historical classification of this malformation consists in four different types, but it is the first one, due to a congenital small posterior fossa, which represent our focus of interest. Chiari malformation may leads to direct brainstem compression and to cerebrospinal fluid circulation trouble at this level, being cause of classical associated phenomena such as syringomyelia formation.

The clinical manifestation may be resumed as follow:

* Exertional headaches or neck pain.
* Brainstem compression signs and symptoms (central apneas syndrome, tetraparesis, paresthesia, cranial nerves disfunction...).
* Syringomyelia signes and symptoms (neuropathic pain, suspended hypo-anesthesia).

The only treatment for Chiari I malformation is the surgical one. It consists in an osteo-dural decompression of the posterior fossa. Surgical decision is formal when at least one of the following criteria is satisfied:

* presence of syringomyelia;
* coexistence of central apneas syndrome;
* presence of the classical symptomatology. Nevertheless, the spectrum of symptoms which might be reported by the patient, and which has even been described in the non neurosurgical literature, is largely wider than the previously thought and assumed by the neurosurgeons. There are so several "atypical symptoms" in which neurosurgeons doesn't believed, and that don't constitute an indicator for surgical intervention. Among these "atypical symptoms" one cas find those ones who bring back to ear, nose and throat domain, such as nystagmus, dizziness, tinnitus, hear loss, and gait instability.

We decided to focalise about one of these symptoms, the gait instability, trying to find the link between Chiari malformation and postural control. In the literature, there are only one study concerning this aspect, conducted on an adult population with the help of a static posturography.

Our study will focus on pediatric patients, who will be evaluated by a dynamic posturography, the Equitest platform (NeuroCom, Clackamas, OR). This platform is able to quantify the contribution of each of the three sensory informations (visual, vestibular and somatosensory) necessary to maintain equilibrium, realising a specific test (Sensory Organisation Test).

The Equitest can elaborate a Composite Equilibrium Score (CES), that will be our PRIMARY JUDGMENT CRITERIA.

Only patients for which ENT evaluation is indicated for medical reasons (for example, children presented frequent falls, dizziness, nystagmus, motion sickness...) will be evaluated.

This evaluation won't change habitual neurosurgical care for the patients presenting Chiari I malformation, so two groups of patients will be identified: children who will be operated on and children who won't. CES of the two groups will be calculated and compared.

Furthermore, we will compared CES results of the operated patients group before and after surgery, to evaluate the impact of surgery on postural control.

In parallel, we will evaluate others SECONDARY CRITERIA in operated patient, before and after surgery, such as :

* signe and symptomss modification;
* decompression result on MRI images;
* syringomyelia modification, if present before;
* central apnea syndrome modification, if present before;
* scoliosis modification, if present before;
* behavioral modification. Anamnestic and clinical data will be part of the habitual computerized medical folder, as well as polysomnographic, posturographic and imaging ones.

Clinical elements of recruited patients will be collected by principal investigator in an anonymous database, secured by a password.

Concerning primary criteria, collected qualitative data will be analysed by Chi-2 or Fischer test, while quantitative ones will be analysed by Student's test or Mann-Whitney one.

Concerning secondary criteria, collected qualitative data will be analysed by Mc Nemar test or symmetry test, while quantitative ones will be analysed by Student's test Wilcoxon one.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically confirmed diagnosis of Chiari I malformation (first MRI realized up to 1/01/2018)
* ENT symptomes (dizziness, nystagmus, gait imbalance, migraines not due to the presence of Chiari Malformation)

Exclusion Criteria:

* Lack of cooperation (cerebral palsy, severe behavioral troubles, orthopedic illness, severe visual impairment)
* Patient's consent for study non obtained.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients aged from 6 to 18 years, received for neurosurgical counseling at our institution with a radiologically confirmed Chiari I malformation and presenting ENT symptomes like dizziness, nystagmus, gait imbalance, motion sickness and Chiari not-related migraines.
  Patients will be selected for surgery in habitual fashion, indipendently on the study.
  The patients will be divided into 2 groups: patients who will be operated on and patients who won't be operated on.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Composite Equilibrium Score | Operated patients: from first neurosurgical evaluation to 6 months after surgery (totally: 8-12 months). Non operated patients: about 4 months for complete evaluation.
  Score elaborated by the Equitest posturography

SECONDARY OUTCOMES:
Cranio cervical MRI | Operated patients: from first neurosurgical evaluation to 6 months after surgery (totally: 8-12 months).
  Posterior fossa decompression
Medullary MRI | Operated patients: from first neurosurgical evaluation to 6 months after surgery (totally: 8-12 months).
  Eventual modification in syringomyelia size
Apnea syndrome | Operated patients: from first evaluation to 6 months after surgery (totally: 8-12 months).
  Eventual modification in polysomnographic results (50% reduction of apnea-hypopnea index)
Clinic | Operated patients: from first neurosurgical evaluation to 6 months after surgery (totally: 8-12 months).
  Eventual modification of patient's signes and symptoms
Scoliosis | Operated patients: from first neurosurgical evaluation to 6 months after surgery (totally: 8-12 months).
  Eventual modification of vertebral balance (favorable outcome if Cobb's angle stable)
Behavior | Operated patients: from first neurosurgical evaluation to 6 months after surgery (totally: 8-12 months).
  Parent's description of behavioral trouble

CONTACTS AND LOCATIONS:
Overall Officials: Perrin Philippe, PhD, Study Director — Nancy Regional University Hospital
Locations (1):
- Stella Irene, Vandœuvre-lès-Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stella I, Remen T, Petel A, Joud A, Klein O, Perrin P. Postural control in Chiari I malformation: protocol for a paediatric prospective, observational cohort - potential role of posturography for surgical indication. BMJ Open. 2022 May 12;12(5):e056647. doi: 10.1136/bmjopen-2021-056647. PMID 35551083